CLINICAL TRIAL: NCT06446128
Title: A Dose Escalating Study of CD19/CD22/BCMA Three Targets Autologous Chimeric Antigen Receptor T (CAR-T) Cell Therapy in Subjects With Relapsed or Refractory B Cell Non-Hodgkin Lymphoma(NHL)
Brief Title: A Dose Escalating Study of CD19/CD22/BCMA CAR-T Therapy in Relapsed or Refractory B Cell Non-Hodgkin Lymphoma(NHL)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Cell Therapy Group Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BZE2204-A-01
Record Dates: First submitted 2024-05-16; First posted 2024-06-06 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Non-Hodgkin Lymphoma, B-cell
Keywords: B cell non-hodgkin lymphoma; CAR-T; CD19; CD22; BCMA
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD19/CD20/BCMA CAR T therapy (Experimental): The safety and tolerability of BZE2204 will be assessed in a "1+1+1+3" and "3+3" dose escalation approach in different B-cell non-hodgkin lymphoma
  Interventions: Biological: CD19/CD20/BCMA CAR T cells

INTERVENTIONS:
Biological: CD19/CD20/BCMA CAR T cells — Subjects will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) for the production of CD19/CD20/BCMA CAR T cells.
  Cyclophosphamide and fludarabine will be given from day-5 to day-3 before the infusion for lymphodepletion. On day0 subjects will receive one dose treatment with CD19/CD20/BCMA CAR T cells by intravenous (IV) injection

SUMMARY:
This is a single arm, open-label, dose escalation clinical study to evaluate the safety and tolerability of autologous chimeric antigen receptor T (CAR-T) cells targeting CD19/CD22/BCMA in patients with relapsed or refractory B cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
This is a single arm, open-label, dose escalation investigator initiated (IIT) study, the primary objective is to evaluate the safety and tolerability of CD19/CD22/BCMA CAR-T therapy in patients with B cell non-Hodgkin lymphoma, and determine the maximum tolerated dose (MTD). For the secondary objectives, pharmacokinetics(PK), survival of CAR-T cells in vivo, pharmacodynamics (PD) and efficacy in R/R B cell NHL will be evaluated.

This study flow comprises of a screening phase( ≤28 days prior to apheresis), apheresis phase (occur upon enrollment, ≤10 days prior to infusion), lymphodepletion phase (from Day -5 to Day -3) ,infusion of CD19/CD22/BCMA CAR-T cells on Day0, DLT assessments phase from Day1 to Day 28 and post-treatment follow-up phase (Day 29 and up to end of the study).

ELIGIBILITY:
Key Inclusion Criteria:

* Patients who are diagnosed with relapsed/refractory B cell non-Hodgkin lymphoma , especially

  * Diffuse Large B Cell Lymphoma, not other specified (DLBCL,NOS),
  * Primary Mediastinal Large B Cell Lymphoma (PMBCL)
  * Transformation Follicular Lymphoma (TFL)
  * High grade B-cell lymphoma(HGBCL)
  * High grade B-cell lymphoma (HGBCL) with MYC(myelocytomatosis oncogene) and BCL2(B-cell lymphoma2) /BCL6 (B-cell lymphoma6) rearrangement
* Refractory diseases are defined as one of the following

  * No response to last line of therapy: i. Progressive disease (PD) as best response to most recent therapy regimen; ii. Stable disease (SD) as best response to most recent therapy regimen
  * Not candidate for autologous stem cell transplant (ASCT) or refractory post-ASCT: i. Disease progression (PD) or relapsed ≤12 months of ASCT (must have biopsy proven recurrence in relapsed individuals) ii. If salvage therapy is given post-ASCT, the individual must have had no response to or relapsed after the last line of therapy
* Individuals must have received adequate prior therapy including at a minimum:

  * anti-CD20 monoclonal antibody unless investigator determines that tumor is CD20-negative and
  * an anthracycline containing chemotherapy regimen
* Immunohistochemical staining shows at least two of B cell surface receptor antigen CD19,CD20, BCMA are positive(including weak, medium and strong positive)
* At least one measurable lesion during the screening based on the recommendation for initial evaluation, staging and response assessment of Hodgkin and non-Hodgkin lymphoma.
* Life expectancy ≥ 12 weeks
* Eastern cooperative oncology group (ECOG) performance status of 0 or 1
* Adequate renal, hepatic, pulmonary and cardiac function defined as:

  * Renal function: Serum creatinine ≤ 1.5 upper limit of normal(ULN), or eGFR ≥ 60 mL/min/1.73m2 [eGFR(estimated glomerular filtration rate)=186×age^-0.203×SCr^-1.154（mg/dl）,female×0.742]
  * Hepatic function: i: Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤ 5 ULN and ii: total bilirubin ≤ 2 ULN, except in individuals with Gilbert syndrome (in Gilbert's syndrome patients, those with total bilirubin ≤ 3 ULN and direct bilirubin ≤ 1.5 ULN can be enrolled).iii: International normalized ratio (INR) or prothrombin time (PT) ≤1.5 ULN Pulmonary: Have the minimum level of pulmonary reserve, defined as ≤ CTCAE (Common Terminology Criteria for Adverse Events) grade 1 dyspnea and the SaO2(oxygen saturation)≥ 91% on room air
  * Cardiac: left ventricular ejection fraction (LVEF) ≥50% determined by echocardiogram(ECG) or multigated acquisition scan (MUGA)
* Adequate bone marrow function, define as:

  * absolute neutrophil count (ANC) ≥1 ×10^9/L
  * absolute lymphocyte count (ALC)≥ 0.5 ×10^9/L
  * Platelets ≥50 ×109/L；
  * Hemoglobulin ≥80 g/L; patients with bone marrow involvement can be enrolled if globulin>60 g/L
* Female of child-bearing age and male participants must agree to use effective contraceptive methods until no CAR-T cells can be detected by PCR(polymerase chain reaction) test.

Key Exclusion Criteria:

* Individuals who have antiCD45 or antiCD3 therapy
* Individuals with detectable cerebrospinal fluid malignant cells, or brain metastases, or with a history of primary or secondary CNS (central nervous system) lymphoma, cerebrospinal fluid malignant cells or brain metastases
* Presence or history of CNS disorder such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement
* History of allogeneic stem cell transplantation
* Any of the following situations:

  • HBsAg/ HBeAg positive; HBeAb/HBcAb positive and HBV(hepatitis B virus) DNA copies above the lower test limit;
* HCV(hepatitis C virus) RNA positive
* HIV(human immunodeficiency virus) positive or treponema pallidum positive
* Presence of active or life-threatening fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management.
* Individuals presence of unstable angina or myocardial infarction within 6 months of screening, or other severe/uncontrolled diseases during the screening (eg. Unstable or uncompensated respiratory, cardiac, hepatic or renal disease)
* Presence of uncontrolled arrhythmia with treatment
* Pregnancy or breastfeeding women

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) | Day0-Day28
  Safety
Maximum tolerated dose (MTD) | Day0-Day28
  Tolerability

SECONDARY OUTCOMES:
Maximum Plasma Concentration(Cmax) | Day0-Day28，Day0-undetectable for CAR positive T cells
  Pharmacokinetics (PK)
Maximum Plasma Concentration Time (Tmax) | Day0-Day28，Day0-undetectable for CAR positive T cells
  Pharmacokinetics (PK)
Area Under Curve (AUC) | Day0-Day28，Day0-undetectable for CAR positive T cells
  Pharmacokinetics(PK)
CAR positive T cells | Day0-Day28，Day0-undetectable for CAR positive T cells
  Pharmacokinetics(PK)
Cytokines ( IL(interleukin)-2, IL-4, IL-6, IL-8, IL-10, IL-15, IFN(interferon)-γ, TNF(tumor necrosis factor)-α and MCP( monocyte chemoattractant protein)-1) | Day0-Day28
  Pharmacodynamics (PD)
Overall survival (OS) | Day28,Month2,Month3,Month6,Month9,Month12,Month18,Month24
  Clinical response assessed by Lugano Response Criteria for non-Hodgkin Lymphoma
Progression-free survival (PFS) | Day28,Month2,Month3,Month6,Month9,Month12,Month18,Month24
  Clinical response assessed by Lugano Response Criteria for non-Hodgkin Lymphoma

CONTACTS AND LOCATIONS:
Overall Officials: Jinxing Lou, Principal Investigator — Shanghai Mengchao Cancer Hospital
Locations (1):
- Mengchao Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No